CLINICAL TRIAL: NCT00150462
Title: A Phase I Study of the Safety and Pharmacokinetics of Escalating Intravenous Doses of the Proteasome Inhibitor PR-171 in Patients With Hematological Malignancies
Brief Title: Safety Study of the Proteasome Inhibitor PR-171 (Carfilzomib for Injection) in Patients With Hematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PX-171-002
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Waldenstrom's Macroglobulinemia; Non-Hodgkin's Lymphoma; Hodgkin's Disease; Multiple Myeloma
Keywords: Hematological; Proteasome; Myeloma; Lymphoma
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Neoplasms, Plasma Cell; Lymphoma | interventions — carfilzomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- CFZ 1.2 mg/m² (Experimental): Participants received carfilzomib (CFZ) 1.2 mg/m² administered by intravenous bolus on Days 1, 2, 8, 9, 15 and 16 in 28-day treatment cycles for up to 12 cycles.
  Interventions: Drug: Carfilzomib
- CFZ 2.4 mg/m² (Experimental): Participants received carfilzomib 2.4 mg/m² administered by intravenous bolus on Days 1, 2, 8, 9, 15 and 16 in 28-day treatment cycles for up to 12 cycles.
  Interventions: Drug: Carfilzomib
- CFZ 4.0 mg/m² (Experimental): Participants received carfilzomib 4.0 mg/m² administered by intravenous bolus on Days 1, 2, 8, 9, 15 and 16 in 28-day treatment cycles for up to 12 cycles.
  Interventions: Drug: Carfilzomib
- CFZ 6.0 mg/m² (Experimental): Participants received carfilzomib 6.0 mg/m² administered by intravenous bolus on Days 1, 2, 8, 9, 15 and 16 in 28-day treatment cycles for up to 12 cycles.
  Interventions: Drug: Carfilzomib
- CFZ 8.4 mg/m² (Experimental): Participants received carfilzomib 8.4 mg/m² administered by intravenous bolus on Days 1, 2, 8, 9, 15 and 16 in 28-day treatment cycles for up to 12 cycles.
  Interventions: Drug: Carfilzomib
- CFZ 11.0 mg/m² (Experimental): Participants received carfilzomib 11.0 mg/m² administered by intravenous bolus on Days 1, 2, 8, 9, 15 and 16 in 28-day treatment cycles for up to 12 cycles.
  Interventions: Drug: Carfilzomib
- CFZ 15.0 mg/m² (Experimental): Participants received carfilzomib 115.0 mg/m² administered by intravenous bolus on Days 1, 2, 8, 9, 15 and 16 in 28-day treatment cycles for up to 12 cycles.
  Interventions: Drug: Carfilzomib
- CFZ 20.0 mg/m² (Experimental): Participants received carfilzomib 20.0 mg/m² administered by intravenous bolus on Days 1, 2, 8, 9, 15 and 16 in 28-day treatment cycles for up to 12 cycles.
  Interventions: Drug: Carfilzomib
- CFZ 27.0 mg/m² (Experimental): Participants received carfilzomib 27.0 mg/m² administered by intravenous bolus on Days 1, 2, 8, 9, 15 and 16 in 28-day treatment cycles for up to 12 cycles.
  Interventions: Drug: Carfilzomib
- CFZ 20/27 mg/m² (Experimental): Participants received carfilzomib 20 mg/m² administered by intravenous bolus on Cycle 1 Days 1, 2, 8, 9, 15 and 16, then 27 mg/m² in all subsequent cycles, for up to 12 cycles.
  Interventions: Drug: Carfilzomib
- CFZ 20/27 mg/m² + DEX (Experimental): Participants received carfilzomib 20 mg/m² administered by intravenous bolus on Cycle 1 Days 1, 2, 8, 9, 15 and 16, then 27 mg/m² in all subsequent cycles, for up to 12 cycles. Participants also received 20 mg dexamethasone (DEX) administered before each dose of carfilzomib (i.e. 40 mg weekly).
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Administered as an IV bolus dose
  Other Names: PR-171; Kyprolis
Drug: Dexamethasone — Administered orally prior to carfilzomib
  Arms: CFZ 20/27 mg/m² + DEX

SUMMARY:
The purpose of this study is to test the safety and tolerability of carfilzomib at different dose levels on hematological cancers such as multiple myeloma, non-Hodgkin's lymphoma, Hodgkin's disease, or Waldenstrom's macroglobulinemia. Carfilzomib is a proteasome inhibitor, an enzyme responsible for degrading a wide variety of cellular proteins.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent in accordance with federal, local, and institutional guidelines
2. Males and females ≥18 years of age
3. Histologically confirmed diagnosis of one of the hematologic malignancies below:

   * Multiple myeloma (MM)
   * Non-Hodgkin's lymphoma (NHL)
   * Waldenström's Macroglobulinemia (WM)
   * Hodgkin's disease (HD)
4. Subjects who are refractory or relapsed following at least two prior therapies
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
6. Adequate cardiovascular function without symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction in the previous six months
7. Adequate hepatic function, with bilirubin < 2.0 times the upper limit of normal, and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) of < 3.0 times the upper limit of normal
8. Total white blood cell (WBC) count ≥ 2,000/mm³, absolute neutrophil count (ANC) ≥ 1000/mm³, hemoglobin ≥ 8.0 g/dL, and platelet count ≥ 50,000/mm³

   * Screening ANC should be independent of granulocyte colony stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) support for ≥ 1 week and of pegylated G-CSF for ≥ 2 weeks)
   * Subjects receiving supportive care including erythropoietin, darbepoetin and/or bisphosphonates can continue to do so, but must be transfusion independent; subjects receiving erythropoietic support must remain on the same dose for the first 28 days of study participation
9. An estimated creatinine clearance of ≥ 30 mL/min, calculated using the formula of Cockroft and Gault
10. Serum creatinine ≤ 2.0 mg/dL
11. Uric acid, if elevated, must be corrected to within laboratory normal range prior to dosing
12. Female subjects of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test. Male subjects must use an effective barrier method of contraception throughout the study and for three months following the last dose if sexually active with a female of child-bearing potential.

Exclusion Criteria:

1. Female subjects who are pregnant or lactating
2. Subjects who are transfusion dependent
3. Subjects with NHL or HL who have received steroid therapy in the previous seven days
4. Subjects with MM or Waldenström's Macroglobulinemia who have received steroid therapy in the previous three weeks, except for MM subjects in the Carfilzomib + DEX Expansion Cohort, where previous treatment with dexamethasone will be allowed. The dose and schedule of administration of dexamethasone will be adjusted to that used in the protocol
5. Radiation, chemotherapy, or immunotherapy in the previous four weeks, or subjects who, in the judgment of the Investigator, have not recovered from the effects of previous therapy
6. For the Dose Escalation period, subjects who have received prior radioimmunotherapy with anti-cluster of differentiation (CD)20 monoclonal antibodies such as Bexxar® or Zevalin®; subjects treated with these products will be allowed in the Dose Expansion period
7. Subjects who have received allogeneic stem cell transplant therapy
8. Subjects with NHL or HL who have received autologous stem cell transplant therapy and have relapsed within 100 days of therapy
9. Rituxan therapy within three months before Day 1 unless there is evidence of disease progression
10. Major surgery within three weeks before Day 1
11. Congestive heart failure (CHF) (New York Heart Association class III to IV)
12. Acute active infection requiring systemic antibiotics, antivirals, or antifungals within two weeks prior to first dose
13. Subjects who are known or suspected of having human immunodeficiency virus (HIV) infection or who are HIV seropositive
14. Active hepatitis A, B, or C infection; or positive for Hepatitis C ribonucleic acid (RNA) or hepatitis B antigen
15. Non-hematologic malignancy within the past three years except a) adequately treated basal cell or squamous cell skin cancer, b) carcinoma in situ of the cervix, or c) prostate cancer with stable prostate specific antigen (PSA) levels for three years
16. Subjects with treatment-related myelodysplastic disorder
17. Subjects with known brain metastasis (active central nervous system [CNS] disease only)
18. Serious psychiatric or medical conditions that could interfere with treatment
19. Participation in an investigational therapeutic study within one month prior to Day 1
20. Significant neurotoxicity (Grade 2 or higher with pain) at the time of study initiation
21. Concurrent therapy with approved or investigative anticancer therapeutics
22. Subjects with previous hypersensitivity to bortezomib injection
23. Subjects with contraindications to receiving allopurinol
24. Subjects in whom the required program of oral and intravenous fluid hydration is contraindicated, e.g., due to pre-existing pulmonary, cardiac, or renal impairment
25. Subjects with known or suspected amyloidosis
26. Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (5):
- United States (5):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weil Medical College of Cornell University, New York, New York
  - Herbert Irving Comprehensive Cancer Center, Columbia University, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults with with multiple myeloma (MM)-both secretory and nonsecretory, non-Hodgkin's lymphoma (NHL), Hodgkin's disease (HD), or Waldenström's macroglobulinemia (WM) were eligible for enrollment in this study.
Pre-assignment Details: The study was divided into a sequential Dose Escalation phase (Part 1; Arms 1-9), followed by a Dose Expansion phase (Part 2; Arms 10-11) consisting of a carfilzomib-only cohort and a carfilzomib-plus dexamethasone cohort.
Groups:
- CFZ 15.0 mg/m²: Participants received carfilzomib 15.0 mg/m² administered by intravenous bolus on Days 1, 2, 8, 9, 15 and 16 in 28-day treatment cycles for up to 12 cycles.
Period: Overall Study
Arm/Group | CFZ 1.2 mg/m² | CFZ 2.4 mg/m² | CFZ 4.0 mg/m² | CFZ 6.0 mg/m² | CFZ 8.4 mg/m² | CFZ 11.0 mg/m² | CFZ 15.0 mg/m² | CFZ 20.0 mg/m² | CFZ 27.0 mg/m² | CFZ 20/27 mg/m² | CFZ 20/27 mg/m² + DEX
Started | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 8 | 6 | 7 | 4
Completed | 0 (Indicates participants remaining on study treatment) | 0 (Indicates participants remaining on study treatment) | 0 (Indicates participants remaining on study treatment) | 0 (Indicates participants remaining on study treatment) | 0 (Indicates participants remaining on study treatment) | 0 (Indicates participants remaining on study treatment) | 0 (Indicates participants remaining on study treatment) | 0 (Indicates participants remaining on study treatment) | 0 (Indicates participants remaining on study treatment) | 1 (Indicates participants who completed 12 cycles of treatment.) | 1 (Indicates participants who completed 12 cycles of treatment.)
Not Completed | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 8 | 6 | 6 | 3
Not completed — Disease Progression or Relapse | 3 | 1 | 2 | 1 | 2 | 2 | 3 | 5 | 5 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CFZ 1.2 mg/m² | CFZ 2.4 mg/m² | CFZ 4.0 mg/m² | CFZ 6.0 mg/m² | CFZ 8.4 mg/m² | CFZ 11.0 mg/m² | CFZ 15.0 mg/m² | CFZ 20.0 mg/m² | CFZ 27.0 mg/m² | CFZ 20/27 mg/m² | CFZ 20/27 mg/m² + DEX | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 8 | 6 | 7 | 4 | 48
Age, Continuous [Mean (Standard Deviation); unit: years]
  Dose Escalation (Part 1) | 62.5 (17.47) | 69.6 (4.80) | 55.3 (21.71) | 51.7 (6.20) | 61.6 (9.15) | 61.3 (3.76) | 50.3 (12.99) | 60.6 (11.99) | 67.6 (9.82) | NA (NA) — Not applicable for Part 2 groups | NA (NA) — Not applicable for Part 2 groups | 60.6 (12.25)
  Dose Expansion (Part 2) | NA (NA) — Not applicable for Part 1 groups | NA (NA) — Not applicable for Part 1 groups | NA (NA) — Not applicable for Part 1 groups | NA (NA) — Not applicable for Part 1 groups | NA (NA) — Not applicable for Part 1 groups | NA (NA) — Not applicable for Part 1 groups | NA (NA) — Not applicable for Part 1 groups | NA (NA) — Not applicable for Part 1 groups | NA (NA) — Not applicable for Part 1 groups | 66.3 (9.21) | 54.3 (13.57) | 61.9 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 3 | 2 | 1 | 4 | 1 | 2 | 2 | 2 | 3 | 22
  Male | 3 | 1 | 1 | 1 | 2 | 0 | 2 | 6 | 4 | 5 | 1 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3
  Caucasian | 3 | 2 | 3 | 3 | 2 | 4 | 3 | 7 | 6 | 6 | 3 | 42
  Hispanic | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Disease Diagnosis [Number; unit: participants]
  Multiple Myeloma | 0 | 3 | 0 | 2 | 1 | 2 | 2 | 6 | 5 | 3 | 4 | 28
  Non-Hodgkin's Lymphoma | 3 | 0 | 3 | 1 | 2 | 2 | 1 | 2 | 1 | 2 | 0 | 17
  Waldenstrom's Macroglobulinemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Hodgkin's Disease | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: A DLT was defined as any of the following occurring in the first 28 days of study participation:
  Nonhematologic:
  * > Grade 2 neuropathy with pain
  * ≥ Grade 3 nonhematologic toxicity (excluding nausea, vomiting, or diarrhea)
  * ≥ Grade 3 nausea, vomiting, or diarrhea uncontrolled by maximal antiemetic/antidiarrheal therapy
  Hematologic:
  * Grade 4 neutropenia (absolute neutrophil count [ANC] < 0.5 × 10ˆ9/L) lasting ≥ 14 days without hematopoietic growth factor support
  * Febrile neutropenia (ANC < 1.0 × 10ˆ9/L with a fever ≥ 38.3°C)
  * Grade 4 thrombocytopenia (platelets < 25.0 × 10ˆ9/L) or thrombocytopenia associated with bleeding.
  Toxicities were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) of the National Cancer Institute (NCI) version 3.0.
Time Frame: 28 days
Population: Safety-evaluable: All participants who were enrolled and received at least 1 dose of carfilzomib
Measure: Number; unit: participants
Arm/Group | CFZ 1.2 mg/m² | CFZ 2.4 mg/m² | CFZ 4.0 mg/m² | CFZ 6.0 mg/m² | CFZ 8.4 mg/m² | CFZ 11.0 mg/m² | CFZ 15.0 mg/m² | CFZ 20.0 mg/m² | CFZ 27.0 mg/m² | CFZ 20/27 mg/m² | CFZ 20/27 mg/m² + DEX
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 8 | 6 | 7 | 4
participants | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1

2. Primary Outcome: Maximum Observed Plasma Concentration of Carfilzomib (Cmax)
Time Frame: Cycle 1, Day 1 at predose, 5, 15, and 30 minutes, and 1, 2, 4, and 24 hours post dose.
Population: Participants with available pharmacokinetic (PK) data. Cmax was only determined for cohorts receiving carfilzomib ≥ 11 mg/m². For cohorts with carfilzomib dose at 1.2-8.4 mg/m², carfilzomib was measurable at too few time points to allow a good estimation. Participants in the two Dose Expansion cohorts (20/27 mg/m²) were combined for PK analyses.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- CFZ 20/27 mg/m² (±DEX): Participants in the Dose Expansion phase received carfilzomib 20 mg/m² administered by intravenous bolus on Cycle 1 Days 1, 2, 8, 9, 15 and 16, then 27 mg/m² in all subsequent cycles, for up to 12 cycles.
Arm/Group | CFZ 1.2 mg/m² | CFZ 2.4 mg/m² | CFZ 4.0 mg/m² | CFZ 6.0 mg/m² | CFZ 8.4 mg/m² | CFZ 11.0 mg/m² | CFZ 15.0 mg/m² | CFZ 20.0 mg/m² | CFZ 27.0 mg/m² | CFZ 20/27 mg/m² (±DEX)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 8 | 5 | 8
ng/mL |  |  |  |  |  | 505.17 (485.12) | 142.67 (97.22) | 527.50 (405.59) | 406.08 (517.29) | 390.66 (492.92)

3. Secondary Outcome: Best Clinical Response to Treatment
Description: Disease response criteria for NHL were according to the International Working Group Criteria for Non-Hodgkin's Lymphoma. Disease response criteria for Multiple Myeloma were according to the European Group for Blood and Marrow Transplantation (EBMT). Disease response criteria for WM were according to the consensus panel recommendations from the Second International Workshop on Waldenström's Macroglobulinemia. The disease response criteria for Hodgkin's Lymphoma are defined as follows:
  * Complete response: total resolution of measurable disease parameters.
  * Partial response: a ≥ 50% resolution without the appearance of new disease.
  * Stable disease: between < 50% resolution and ≤ 25% increases in measurable disease parameters without appearance of new disease.
  * Progressive disease: an increase of > 25% in measurable disease parameters.
  Best clinical response is the best response observed from the start of study treatment until disease progression or death.
Time Frame: From the first dose of study drug until 30 days after the last dose. Median duration of treatment was 6.3 weeks in the dose escalation phase and 6.4 weeks in the dose expansion phase.
Population: Biologic response-evaluable: All participants who received at least 1 cycle of carfilzomib and had both baseline and at least 1 post-baseline disease assessment.
Measure: Number; unit: participants
Arm/Group | CFZ 1.2 mg/m² | CFZ 2.4 mg/m² | CFZ 4.0 mg/m² | CFZ 6.0 mg/m² | CFZ 8.4 mg/m² | CFZ 11.0 mg/m² | CFZ 15.0 mg/m² | CFZ 20.0 mg/m² | CFZ 27.0 mg/m² | CFZ 20/27 mg/m² | CFZ 20/27 mg/m² + DEX
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 3 | 3 | 2 | 6 | 5 | 6 | 3
participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 0
  Minimal Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Stable Disease/No Change | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 2 | 1 | 2 | 0
  Progressive Disease | 1 | 1 | 1 | 0 | 2 | 2 | 1 | 3 | 1 | 2 | 2
  Unknown | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Duration of Response
Description: Duration of objective response is defined as the time from the date of first documented assessment of clinical response (confirmed or unconfirmed complete response, partial response, or minimal response) to the date of documented assessment of progressive disease or death, whichever comes first, plus one day. Participants without tumor progression or death were censored at the date of their last valid clinical response assessment.
  Median duration of response was calculated using the Kaplan-Meier method.
Time Frame: as for outcome 3
Population: Biologic response-evaluable participants with an objective response
Measure: Median (Full Range); unit: days
Groups:
- CFZ 20/27 mg/m²: Participants received carfilzomib 20 mg/m² administered by intravenous bolus on Cycle 1 Days 1, 2, 8, 9, 15, and 16, then 27 mg/m² in all subsequent cycles, for up to 12 cycles.
- CFZ 20/27 mg/m² + DEX: Participants received carfilzomib 20 mg/m² administered by intravenous bolus on Cycle 1 Days 1, 2, 8, 9, 15, and 16, then 27 mg/m² in all subsequent cycles, for up to 12 cycles. Participants also received 20 mg dexamethasone (DEX) administered before each dose of carfilzomib (i.e. 40 mg weekly).
Arm/Group | CFZ 1.2 mg/m² | CFZ 2.4 mg/m² | CFZ 4.0 mg/m² | CFZ 6.0 mg/m² | CFZ 8.4 mg/m² | CFZ 11.0 mg/m² | CFZ 15.0 mg/m² | CFZ 20.0 mg/m² | CFZ 27.0 mg/m² | CFZ 20/27 mg/m² | CFZ 20/27 mg/m² + DEX
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 2 | 1
days |  |  |  |  |  |  | 308.0 [308.0 to 308.0] | 176.0 [176.0 to 176.0] | 225.0 [94.0 to 316.0] | NA [NA to NA] — Could not be calculated due to the low number of events | NA [NA to NA] — Could not be calculated due to the low number of events

5. Secondary Outcome: Time to Progression
Description: Time to progressive disease is defined as the time from the date of Cycle 1, Day 1 of treatment to the date of documented assessment of progressive disease, plus one day. Participants without tumor progression were censored at the date of their last clinical response assessment.
  Median time to progression was calculated using the Kaplan-Meier method.
Time Frame: as for outcome 3
Population: Biologic response-evaluable population
Measure: Median (Full Range); unit: days
Arm/Group | CFZ 1.2 mg/m² | CFZ 2.4 mg/m² | CFZ 4.0 mg/m² | CFZ 6.0 mg/m² | CFZ 8.4 mg/m² | CFZ 11.0 mg/m² | CFZ 15.0 mg/m² | CFZ 20.0 mg/m² | CFZ 27.0 mg/m² | CFZ 20/27 mg/m² | CFZ 20/27 mg/m² + DEX
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 3 | 3 | 2 | 6 | 5 | 6 | 3
days | 114.0 [114.0 to 114.0] | 232.0 [57.0 to 407.0] | NA [54.0 to 54.0] — Not estimable due to the low number of events | NA [NA to NA] — Not estimable due to the low number of events | 55.0 [47.0 to 55.0] | 48.0 [15.0 to 176.0] | 186.0 [50.0 to 322.0] | 110.5 [15.0 to 190.0] | 225.0 [36.0 to 330.0] | NA [15.0 to 99.0] — Not estimable due to the low number of events | 49.0 [23.0 to 49.0]

6. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from the date of Cycle 1, Day 1 of treatment to the date of documented assessment of progressive disease or death, whichever comes first, plus one day. Participants without tumor progression or death were censored at the date of their last valid clinical response assessment. Median progression-free survival was calculated using the Kaplan-Meier method.
Time Frame: as for outcome 3
Population: Biologic response-evaluable population
Measure: Median (Full Range); unit: days
Arm/Group | CFZ 1.2 mg/m² | CFZ 2.4 mg/m² | CFZ 4.0 mg/m² | CFZ 6.0 mg/m² | CFZ 8.4 mg/m² | CFZ 11.0 mg/m² | CFZ 15.0 mg/m² | CFZ 20.0 mg/m² | CFZ 27.0 mg/m² | CFZ 20/27 mg/m² | CFZ 20/27 mg/m² + DEX
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 3 | 3 | 2 | 6 | 5 | 6 | 3
days | 114.0 [114.0 to 114.0] | 232.0 [57.0 to 407.0] | NA [54.0 to 54.0] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | 55.0 [47.0 to 55.0] | 48.0 [15.0 to 176.0] | 186.0 [50.0 to 322.0] | 110.5 [15.0 to 190.0] | 225.0 [36.0 to 330.0] | NA [15.0 to 99.0] — Could not be estimated due to the low number of events | 49.0 [23.0 to 49.0]

7. Primary Outcome: Time to Maximum Observed Plasma Concentration of Carfilzomib (Tmax)
Time Frame: Cycle 1, Day 1 at predose, 5, 15, and 30 minutes, and 1, 2, 4, and 24 hours post dose.
Population: Participants with available pharmacokinetic (PK) data. Tmax was only determined for cohorts receiving carfilzomib ≥ 11 mg/m². For cohorts with carfilzomib dose at 1.2-8.4 mg/m², carfilzomib was measurable at too few time points to allow a good estimation. Participants in the two Dose Expansion cohorts (20/27 mg/m²) were combined for PK analyses.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | CFZ 1.2 mg/m² | CFZ 2.4 mg/m² | CFZ 4.0 mg/m² | CFZ 6.0 mg/m² | CFZ 8.4 mg/m² | CFZ 11.0 mg/m² | CFZ 15.0 mg/m² | CFZ 20.0 mg/m² | CFZ 27.0 mg/m² | CFZ 20/27 mg/m² (±DEX)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 8 | 5 | 8
minutes |  |  |  |  |  | 5 (0) | 6 (1) | 7 (2) | 6 (2) | 16 (11)

8. Primary Outcome: Area Under the Concentration-time Curve to Last Measureable Timepoint (AUClast) for Carfilzomib
Time Frame: Cycle 1, Day 1 at predose, 5, 15, and 30 minutes, and 1, 2, 4, and 24 hours post dose.
Population: Participants with available pharmacokinetic (PK) data. AUClast was only determined for cohorts receiving carfilzomib ≥ 11 mg/m². For cohorts with carfilzomib dose at 1.2-8.4 mg/m², carfilzomib was measurable at too few time points to allow a good estimation. Participants in the two Dose Expansion cohorts (20/27 mg/m²) were combined for PK analyses.
Measure: Mean (Standard Deviation); unit: ng*minute/mL
Arm/Group | CFZ 1.2 mg/m² | CFZ 2.4 mg/m² | CFZ 4.0 mg/m² | CFZ 6.0 mg/m² | CFZ 8.4 mg/m² | CFZ 11.0 mg/m² | CFZ 15.0 mg/m² | CFZ 20.0 mg/m² | CFZ 27.0 mg/m² | CFZ 20/27 mg/m² (±DEX)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 8 | 5 | 8
ng*minute/mL |  |  |  |  |  | 4049 (3695) | 1414 (919) | 4911 (3495) | 3409 (3964) | 4970 (5817)

9. Primary Outcome: Area Under the Concentration-time Curve Extrapolated to Infinity (AUCinf) for Carfilzomib
Time Frame: Cycle 1, Day 1 at predose, 5, 15, and 30 minutes, and 1, 2, 4, and 24 hours post dose.
Population: Participants with available pharmacokinetic (PK) data. AUCinf was only determined for cohorts receiving carfilzomib ≥ 11 mg/m². For cohorts with carfilzomib dose at 1.2-8.4 mg/m², carfilzomib was measurable at too few time points to allow a good estimation. Participants in the two Dose Expansion cohorts (20/27 mg/m²) were combined for PK analyses.
Measure: Mean (Standard Deviation); unit: ng*minute/mL
Arm/Group | CFZ 1.2 mg/m² | CFZ 2.4 mg/m² | CFZ 4.0 mg/m² | CFZ 6.0 mg/m² | CFZ 8.4 mg/m² | CFZ 11.0 mg/m² | CFZ 15.0 mg/m² | CFZ 20.0 mg/m² | CFZ 27.0 mg/m² | CFZ 20/27 mg/m² (±DEX)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 8 | 5 | 8
ng*minute/mL |  |  |  |  |  | 4056 (3698) | 1420 (922) | 4942 (3497) | 3417 (3962) | 4997 (5812)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 30 days after the last dose. Median duration of treatment was 6.3 weeks in the dose escalation phase and 6.4 weeks in the dose expansion phase.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | CFZ 1.2 mg/m² | CFZ 2.4 mg/m² | CFZ 4.0 mg/m² | CFZ 6.0 mg/m² | CFZ 8.4 mg/m² | CFZ 11.0 mg/m² | CFZ 15.0 mg/m² | CFZ 20.0 mg/m² | CFZ 27.0 mg/m² | CFZ 20/27 mg/m² | CFZ 20/27 mg/m² + DEX
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 3/4 | 2/3 | 2/3 | 2/4 | 1/3 | 3/8 | 4/6 | 3/7 | 2/4
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 3/3 | 3/3 | 4/4 | 3/3 | 8/8 | 6/6 | 7/7 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CFZ 1.2 mg/m² (N=3) | CFZ 2.4 mg/m² (N=3) | CFZ 4.0 mg/m² (N=4) | CFZ 6.0 mg/m² (N=3) | CFZ 8.4 mg/m² (N=3) | CFZ 11.0 mg/m² (N=4) | CFZ 15.0 mg/m² (N=3) | CFZ 20.0 mg/m² (N=8) | CFZ 27.0 mg/m² (N=6) | CFZ 20/27 mg/m² (N=7) | CFZ 20/27 mg/m² + DEX (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Unresponsive to verbal stimuli (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CFZ 1.2 mg/m² (N=3) | CFZ 2.4 mg/m² (N=3) | CFZ 4.0 mg/m² (N=4) | CFZ 6.0 mg/m² (N=3) | CFZ 8.4 mg/m² (N=3) | CFZ 11.0 mg/m² (N=4) | CFZ 15.0 mg/m² (N=3) | CFZ 20.0 mg/m² (N=8) | CFZ 27.0 mg/m² (N=6) | CFZ 20/27 mg/m² (N=7) | CFZ 20/27 mg/m² + DEX (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 2 | 0 | 1 | 2 | 4 | 4 | 4 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 3 | 3 | 4 | 3
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Exophthalmos (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 2 | 1 | 2 | 2 | 0 | 4 | 3 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 1 | 2 | 0 | 2 | 2 | 3 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 3 | 1 | 2 | 2 | 3 | 5 | 4 | 3 | 0
Oedema mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 2 | 1 | 3 | 1 | 2 | 1 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 2 | 2 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 3 | 1 | 1 | 3 | 3 | 3 | 3 | 4 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Infusion site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 3 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Pitting oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 3 | 0 | 1 | 1 | 2 | 2 | 3 | 3 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Echinococciasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial natriuretic peptide increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 3 | 3 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 4 | 1 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 5 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 3 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asterixis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 2 | 1 | 2 | 1 | 0 | 2 | 2 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 3 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 3 | 1
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bladder disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 3 | 2 | 1 | 0 | 4 | 3 | 1
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 4 | 2 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal sinus drainage (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.